CLINICAL TRIAL: NCT02517840
Title: Revascularization Results in Nonagenarian Patients With Critical Lower Limb Ischaemia
Brief Title: Revascularization in Nonagenarian Patients With Critical Lower Limb Ischaemia
Acronym: NONA-CLI
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, Joaquin de Haro, M.D., Joaquin de Haro, M.D., Hospital Universitario Getafe
Other Study IDs: 15/199 ESTUDIO
Record Dates: First submitted 2015-07-26; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nonagenarian CLI: Patients suffering from Critical Limb Ischemia aged 90 year-old or above who undergo limb revascularization by means of open surgery or endovascular revascularization

SUMMARY:
The rise in life expectancy implies an increased number of nonagenarian patients who need evaluation for critical lower limb ischaemia (CLI). The study goal is to evaluate whether revascularization techniques in these patients fulfill a set of security and efficacy criteria generated from surgical results in a validated historical cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Critical Limb Ischemia aged 90 year-old or above

Exclusion Criteria:

-

Min Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients suffering from Critical Limb Ischemia aged 90 year-old or above
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2002-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence at 30 days of major adverse cardiovascular events (MACE) | 30 days after the procedure
  Incidence at 30 days of major adverse cardiovascular events (MACE): stroke, myocardial infarction or death by cardiovascular cause, in percentage.
Incidence at 30 days of major adverse limb events (MALE) | 30 days after the procedure
  Incidence at 30 days of major adverse limb events (MALE): limb acute ischemia or amputation, in percentage.
Incidence at 30 days of limb major amputations (MA) | 30 days after the procedure
  Incidence at 30 days of limb major amputations (MA), in percentage.

SECONDARY OUTCOMES:
Limb salvage (LS) | 12 months after the procedure
  Percentage of revascularized limb which do no require major amputation at 12 months
Survival | 12 months after the procedure
  Percentage of patients alive at 12 months